CLINICAL TRIAL: NCT06878131
Title: Precision-MRD: Prospective Observational Study of Biomarker-directed Systemic Therapy for Colorectal Cancer Patients With Minimal Residual Disease
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-1886
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Colorectal Cancer — Participants that take part in this research, will be responsible for following study directions and allowing blood samples to be collected every 3 months for correlative studies.

SUMMARY:
The goal of this clinical research study is to learn about the effects of biomarkertargeted therapy on ctDNA in patrticipants with CRC and MRD.

This is an observational study. Participants will be monitored while receiving biomarker-directed therapy that is determined by your treating oncologist (cancer doctor) per standard of care, independent of this study.

DETAILED DESCRIPTION:
Primary Objective

• To estimate the rate of ctDNA clearance at 6 months following initiation of biomarker-directed targeted therapy in colorectal cancer (CRC) participants with minimal residual disease (MRD).

Secondary Objectives

* To evaluate dynamics of ctDNA mutant allele fractions following initiation of biomarker-directed targeted therapy in MRD-positive CRC participants.
* To estimate the rate of disease recurrence at 1 year following initiation of biomarker-directed targeted therapy in MRD-positive CRC participants.

ELIGIBILITY:
Inclusion Criteria

1. Male or female subjects aged > 18 years.
2. Histologically or cytologically confirmed diagnosis of colorectal adenocarcinoma.
3. Stage II-IV disease per current AJCC staging criteria with no definitive radiographic evidence of disease following locoregional treatment. Small indeterminate lesions measuring < 10 mm may be permitted at the discretion of the principal investigator.
4. Presence of one of the following targetable biomarkers on tumor or blood molecular testing: BRAF V600E mutation (Cohort A), KRAS G12C mutation (Cohort B), MSI-H status (Cohort C), and HER2 amplification (Cohort D).
5. Positive ctDNA blood test obtained > 21 days after surgery or last administration of adjuvant therapy.
6. Prescribed one of the following standard-of-care targeted therapy regimens: BRAF V600E Inhibitor + anti-EGFR antibody for BRAF V600E-mutated tumors, KRAS G12C Inhibitor + anti-EGFR antibody for KRAS G12C-mutated tumors, anti-PD-1 antibody +/- anti-CTLA-4 antibody for MMRd/MSI-H tumors, or anti-HER2 therapies for HER2 amplified tumors.

Exclusion Criteria

1. Prior exposure to the following classes of biomarker-directed therapies: BRAF V600E inhibitors, anti-EGFR antibodies, KRAS G12C inhibitors, anti-PD-1/PD-L1 antibodies, anti-CTLA-4 antibodies, or anti-HER2 therapies
2. Presence of a concurrent malignancy requiring active treatment
3. Inability to provide informed consent
4. Children will not be enrolled in this study
5. Pregnant women will not be enrolled in this study
6. Cognitively Impaired subjects will not be enrolled in this study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: MD Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-04-18 (Actual); Primary Completion 2026-12-22 (Estimated); Study Completion 2028-12-22 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse events (AEs) | Through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Saurav Haldar, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: Related Info — http://www.mdanderson.org